CLINICAL TRIAL: NCT05175794
Title: Phase 4 Operational Study to Assess the Effectiveness, Feasibility, Acceptability, and Cost-effectiveness of the GeneXpert MTB/XDR (Xpert XDR; Cepheid) Assay for Rapid Triage-and-treatment of DR-TB
Brief Title: Triage Test for All Oral DR-TB Regimen (TRiAD Study)
Status: Completed | Type: Observational
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: KNCV Tuberculosis Foundation (Other); Amsterdam Institute for Global Health and Development (Other); Ospedale San Raffaele (Other); Foundation for Innovative New Diagnostics, Switzerland (Other); National Institute for Medical Research, Tanzania (Other Government); University of St Andrews (Other); Global Alliance for TB Drug Development (Other); Wits Health Consortium (Pty) Ltd (Other); Institute of Human Virology, Nigeria (Other); Ethiopian Public Health Institute (Other Government)
Responsible Party: Principal Investigator, Dr Kogieleum Naidoo, Associate Professor, Centre for the AIDS Programme of Research in South Africa
Other Study IDs: CAPRISA 094; TRIAD (Other: CAPRISA)
Record Dates: First submitted 2021-09-22; First posted 2022-01-04 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Drug Resistant Tuberculosis; MDR-TB; XDR-TB; Tuberculosis
Keywords: GeneXpert; Diagnostic Tool
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to provide sputum samples for this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants that test positive for Mycobacterium tuberculosis (M.tb) with rifampicin resistance will be enrolled in Cohort 1 (n=880).
  Interventions: Diagnostic Test: Xpert® MTB/XDR
- Cohort 2: Participants that test positive for M.tb that are rifampicin susceptible with isoniazid mono-resistance will be enrolled in Cohort 2 (n=400).
  Interventions: Diagnostic Test: Xpert® MTB/XDR

INTERVENTIONS:
Diagnostic Test: Xpert® MTB/XDR — The Xpert MTB/XDR Assay, performed on the GeneXpert Instrument Systems, is a nested real-time polymerase chain reaction(PCR) in vitro diagnostic test for the detection of extensively drug resistant (XDR) Mycobacterium tuberculosis (MTB) complex DNA in unprocessed sputum samples or concentrated sediments prepared from sputum. In specimens where MTB is detected, the Xpert MTB/XDR Assay can also detect isoniazid (INH) resistance associated mutations in the katG and fabG1 genes, oxyRahpC intergenic region and inhA promoter; ethionamide (ETH) resistance associated with inhA promoter mutations only; fluoroquinolone (FLQ) resistance associated mutations in the gyrA and gyrB quinolone resistance determining regions (QRDR); and second line injectable drug (SLID) associated mutations in the rrs gene and the eis promoter region.
  Other Names: Xpert MTB/XDR Assay; Xpert XDR

SUMMARY:
A Phase 4 operational study to assess the effectiveness, feasibility, acceptability, and cost effectiveness of the GeneXpert MTB/XDR (Xpert XDR; Cepheid) assay for rapid triage-and-treatment of DR-TB-A multi-centre, multi-country prospective cohort study

DETAILED DESCRIPTION:
The TriAD study is a multi-center, multi-country Prospective Pragmatic Cohort study assessing the effectiveness, feasibility, acceptability, and cost-effectiveness of implementing the Xpert MTB/XDR (Xpert XDR; Cepheid) assay for rapid triage-and-treatment with short, all- oral drug resistant tuberculosis (DR-TB) treatment. The proposed study aims to screen approximately 4800 GeneXpert MTB/RIF or Ultra MTB-positive (irrespective of rifampicin resistance status) patients from 9 study sites in South Africa, Nigeria and Ethiopia to enrol 880 rifampicin resistant (RR) and 400 isoniazid mono-resistant (HR) patients over a period of 12-18 months. The Xpert XDR assay, a rapid genotypic test, will be implemented as a reflex test to detect resistance to isoniazid, fluoroquinolones and second-line injectable agents to provide rapid genotypic susceptibility testing for DR-TB detection. Patients that test positive for Mycobacterium tuberculosis with rifampicin resistance will be enrolled in Cohort 1 (n=880). Patients that test positive for Mycobacterium tuberculosis that are rifampicin susceptible with isoniazid mono-resistance will be enrolled in Cohort 2 (n=400). Results from the Xpert XDR assay will be used to guide selection of appropriate, evidence-based, all-oral DR-TB treatment regimens of shortest possible duration. The tuberculosis molecular bacterial load assay (TB-MBLA) will be used as an adjunct to provide bacillary load monitoring over the course of treatment to assess real-time treatment response. Operational research will provide information about the feasibility, acceptability and cost-effectiveness to inform policies and guidelines for programmatic implementation of the triage-and-treat model.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulant adults ≥ 18 years of age
2. Newly diagnosed PTB patients receiving less than 5 days of treatment since new diagnosis:

   1. Cohort 1: < 5 days of DR-TB treatment
   2. Cohort 2: < 5 days of INH mono-resistant TB treatment preceding study entry for the current TB episode, or
3. Sputum positive (smear and or culture) TB patients classified as failing first line treatment
4. Any currently available Nucleic Acid Amplification Tests for drug-resistance detection changes/assay positive for M.tb infection with:

   Cohort 1: at least Rifampicin resistance Cohort 2: Rifampicin susceptible co-occurring with INH, fluoroquinolone, ethionamide or aminoglycoside resistance (detected by Xpert XDR) occurring alone or in combination
5. Capacity to provide informed consent
6. HIV infected and uninfected participants are allowed in the study. Participants already on ART will be allowed in the study provided the ART regimen in use has no contraindications to the proposed TB drug regimen
7. Willing to have samples collected, stored indefinitely, and used for research purposes
8. Able to provide reasonable proof of identity (to satisfaction of study team member) at or prior to enrolment

Exclusion criteria:

1. Has a known severe allergy to any of the BPaL component drugs
2. Has DST showing infection with a strain resistant to any of the component drugs
3. Has TB meningitis, other central nervous system TB, or TB osteomyelitis; or
4. Is pregnant or breastfeeding
5. Is unable to take oral medications
6. Persons with any other medical condition, precluding study participation based on investigator judgement
7. Any co-existing condition that in the opinion of the attending clinician renders the participant unsuitable for participation in the study
8. Co-enrolment in other interventional research studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two screening strategies will be adopted:
  1. Patients with suspected pulmonary TB or confirmed M.tb positive (< 5 days since treatment initiation) will be screened and consented to provide an additional sputum sample for Xpert MTB/XDR testing. This will be in addition to the routine sample collected for GeneXpert MTB/RIF or Ultra testing
  2. We will concurrently contact all patients with newly identified RR-TB during the study enrolment period directly for participation in this study (laboratory records)
Sampling Method: Non-Probability Sample
Enrollment: 786 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Time to initiation | 4 years
  Time to initiation of an appropriate all oral treatment regimen from date of first sputum collected
Proportion of patients with favorable treatment outcomes | 4 years
  Proportion of patients with favorable treatment outcomes at month 12 from diagnosis

SECONDARY OUTCOMES:
Adverse Drug Reactions | 4 years
  Incidence of adverse drug reactions documented during all oral treatment
Mortality | 4 years
  All cause mortality documented during treatment and follow up
Time to culture Conversion | 4 years
  Time specific rates of culture conversion
HR TB Prevalence | 4 years
  Prevalence of HR TB (cohort 2)
XDR TB Prevalence | 4 years
  Prevalence of XDR TB (cohort 2)
Proportion of patients with Bedaquiline and linezolid resistance not eligible for short course treatment | 4 years
  Proportion of patients with Bedaquiline and linezolid resistance not eligible for short course treatment
Clinical utility of the Tuberculosis Molecular Bacterial Load Assay (TB-MBLA) compared to routine culture to monitor DR-TB treatment response | 4 years
  Quantitative results from the TB-MBLA, a real-time quantitative PCR (RT-qPCR) assay, that detects and quantifies killing of 16S rRNA from both viable replicating and dormant M. tuberculosis in patient sputum during treatment, will be compared to routine culture in monitoring treatment response
Feasibility of Tuberculosis Molecular Bacterial Load Assay (TB-MBLA) will be compared to routine culture in bacteriological follow-up for people on DR-TB treatment | 4 years
  Feasibility of TB-MBLA Assessed by comparison to liquid culture with respect to accuracy, result turn-around time, failure rates.
Accuracy of Xpert XDR testing compared to WGS | 4 years
  The performance of Xpert XDR will be compared to Culture DST, LPA and Next Generation Sequencing.
Quality of Xpert XDR testing | 4 years
  Quality of Xpert XDR testing will be assessed using:
  1. indeterminate rates measured by the number of Xpert XDR tests regarded as invalid divided by the total number of Xpert XDR tests performed
  2. Contamination rates or frequency of DNA contamination: number of Xpert XDR tests flagging contamination divided by the total number of Xpert XDR tests performed or events
  3. performance variation will be measured by performance in discrimination of (i) INH resistance compared to culture across study sites, (ii) aminoglycoside resistance compared to culture across study sites and (iii) fluroquinolone resistance compared to culture across study sites
Resistance profile of sputum samples for identification of drug resistance mutations as per pre-existing probes within the Xpert XDR assay | 4 years
  Cultured isolates from the same sputum sample will undergo WGS sequencing to identify additional resistance mutations to new and re-purposed drugs. The endpoints measured for this objective includes:
  1. Frequency of detection of additional resistance conferring mutations by WGS not detected by Xpert XDR
  2. Impact of these previously undetected mutation on conferring resistance to the new drugs in the bedaquiline, pretomanid and linezolid regimen
Cost effectiveness | 4 years
  Data for Costing studies will be collected through semi-structured interviews of key informants and document review. Methods will include a construction of incremental cost effectiveness ratios (ICER) and CE-model to estimate the costs and benefits from a societal perspective, generalizable to other settings.
  timely initiated on treatment
Operational Feasibility of patient triaging | 4 years
  The Operational Cost including Infrastructure and Human resource requirements for the study approach.

CONTACTS AND LOCATIONS:
Overall Officials: Kogieleum Naidoo, MBCHB, PHD, Principal Investigator — Deputy Director -CAPRISA
Locations (4):
- Ethiopian Public Health Institute (EPHI), Gulele, Addis Ababa, Ethiopia
- Institute of Human Virology Nigeria, Yaba, Lagos, Nigeria
- South Africa (2):
  - CAPRISA Springfield Research Clinic, Durban, KwaZulu-Natal
  - Clinical HIV Research Unit (CHRU), WITS Health Consortium, Bethelsdorp, Port Elizabeth

REFERENCES:
- [Background] Conradie F, Diacon AH, Ngubane N, Howell P, Everitt D, Crook AM, Mendel CM, Egizi E, Moreira J, Timm J, McHugh TD, Wills GH, Bateson A, Hunt R, Van Niekerk C, Li M, Olugbosi M, Spigelman M; Nix-TB Trial Team. Treatment of Highly Drug-Resistant Pulmonary Tuberculosis. N Engl J Med. 2020 Mar 5;382(10):893-902. doi: 10.1056/NEJMoa1901814. PMID 32130813
- [Background] Gillespie SH, Sabiiti W, Oravcova K. Mycobacterial Load Assay. Methods Mol Biol. 2017;1616:89-105. doi: 10.1007/978-1-4939-7037-7_5. PMID 28600763
- [Derived] Naidoo K, Naidoo A, Abimiku AG, Tiemersma EW, Gebhard A, Hermans SM, Sloan DJ, Ruhwald M, Georghiou SB, Okpokoro E, Agbaje A, Yae K, Tollera G, Moga S, Feyt H, Kachoka T, Letsoalo MP, Cabibbe AM, Perumal R, Shunmugam L, Cirillo DM, Foraida S, Sabiiti W, Ntinginya NE, Mtafya B, Bedru A, Gillespie SH; TRiAD Study Consortium. Triage test for all-oral drug-resistant tuberculosis (DR-TB) regimen: a phase IV study to assess effectiveness, feasibility, acceptability and cost-effectiveness of the Xpert MTB/XDR assay for rapid triage and treatment of DR-TB. BMJ Open. 2024 Nov 27;14(11):e084722. doi: 10.1136/bmjopen-2024-084722. PMID 39609025
- See also: WHO consolidated guidelines on tuberculosis — http://www.ncbi.nlm.nih.gov/books/NBK572344/

DOCUMENTS (1):
  • Study Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT05175794/Prot_001.pdf